Version

COMIRB
Approved for
RECONSENT
20-Jun-2025
19-Dec-2025

# Optional LUMBAR PUNCTURE Informed Consent and Author Form

STUDY TITLE: Phase II Trial to Evaluate Safety and Efficacy of GM-

CSF/Sargramostim in Alzheimer's Disease (SESAD)

PROTOCOL NUMBER: COMIRB #19-2727

STUDY DRUG: Sargramostim (also referred to as "study drug")

SPONSOR/PRINCIPAL Huntington Potter, PhD INVESTIGATOR: University of Colorado

Alzheimer's and Cognition Center

Mail Stop 8680 12700 E. 19<sup>th</sup> Ave. Aurora, CO 80045

STUDY SITE INFORMATION: University of Colorado

**Anschutz Medical Campus** 

Aurora, CO 80045



#### INTRODUCTION

You are being asked to have optional lumbar puncture as part of the clinical research study Phase II Trial to Evaluate Safety and Efficacy of GM-CSF/Sargramostim in Alzheimer's Disease (SESAD). To help you decide, you should understand the procedure and what it will involve to participate. This form provides you with information about the procedure. A member of the research team will describe this procedure to you and answer all of your questions. Please read the information below and ask questions about anything you don't understand before deciding whether or not to take part.

Some people in this study may have a medical condition or a disability that does not allow them to make important decisions for themselves. If you have been asked to decide for someone else whether they should be in this study, please read this consent form carefully. In this form, we use the words "you" and "your." If you are reading this form and deciding for someone else, the words 'you' and 'your' refer to that other person, not to you.

#### WHY IS THIS OPTIONAL LUMBAR PUNCTURE BEING DONE?

You are being asked to have an optional lumbar puncture because you have been diagnosed with mild-to-moderate Alzheimer's Disease (AD) and have agreed to take part in the Phase II Trial to Evaluate Safety and Efficacy of GM-CSF/Sargramostim in Alzheimer's Disease (SESAD). While **it is** 

**not necessary** to have this lumbar puncture to participate in the main study, as you have chosen to have the Amyloid PET scan for study entry criteria, the lumbar puncture is very valuable for research into the deposition of amyloid beta and tau proteins within the brain, and to give further information to study researchers on what impact, if any, sargramostim has upon these proteins within the brain, as well as other measures of brain health.

#### WHAT WILL HAPPEN IF I HAVE LUMBAR PUNCTURES?

If you consent to participate in the optional lumbar puncture research part of the study, you will receive 2 lumbar puncture procedures in total in the study (1 in the screening portion of the study after the amyloid PET scan visit, and 1 at the End of Treatment visit). It is expected that approximately one-half of participants will take part in the optional lumbar puncture research part of the study. Each lumbar puncture visit should take approximately 1 to 1.5 hours, while the procedure itself should take approximately 30-40 minutes.

Before the lumbar puncture, an experienced clinician will assess your vital signs, and assess you to determine the appropriateness of the procedure. You will either sit on a special chair, or lay on a bed, based upon the judgement of the clinician. The clinician will insert a small needle into your lower back, into your spinal canal, under sterile conditions. The clinician will use an atraumatic needle, designed to reduce the risk of post procedure headache, and collect approximately 25-30 mL (about 2 tablespoons) of cerebrospinal fluid (CSF). This CSF will be used to measure a variety of important markers of Alzheimer's disease progression. After the procedure, you will rest for 30 minutes.

As the results of the optional LP are for research purposes, you will NOT be informed of the results of the test.

#### WHAT ARE THE POSSIBLE DISCOMFORTS OR RISKS?

#### Possible risks of lumbar puncture

Risks associated with lumbar puncture (LP) include pain and/or bleeding at the site of needle insertion. To improve your comfort, the skin, surrounding tissue and underlying muscle will be numbed with a drug called lidocaine. This is similar to the numbing medication delivered during a dental procedure, such as a tooth extraction. Lidocaine injection may cause a burning sensation. This sensation is brief and generally associated only with the administration of the drug. There is also some risk of infection any time the skin is pierced with a needle.

During the LP you may experience brief pain lasting seconds in the lower back during insertion of the needle, especially if the needle contacts bone. This occurs about 1 in 5 times. Less than 1 in 10 patients experience a brief pain shooting down the leg if the LP needle touches a nerve root. Rarely, this sensation or some numbness in the leg may persist for days. Fewer than 1 in 100 patients are allergic to the iodine solution used to clean their back and will develop rash.

After an LP, about 10 out of 100 individuals may develop a headache, which is typically mild. It typically begins 6-48 hours after the LP, and may last 1 to 6 days. Lying flat, staying well hydrated, and taking caffeine (not provided by the study) usually helps the headache to resolve. To reduce the likelihood of a temporary headache after the LP, you may be asked to rest for a short period of time after the procedure. Post-LP headache may be treated with oral hydration, analgesics such as

acetaminophen, or ibuprofen and caffeine (not provided by the study). We will also call you the day after your spinal fluid collection to see how you are feeling.

A more severe headache can occur after a lumbar puncture, but it is rare. To minimize risk, we use a special type of needle (called an atraumatic needle) in all of our research studies. With this type of special needle, the risk of a severe headache has been shown to be very low –approximately 1% or less. These types of headaches are typically responsive to treatment within a few hours. If the severe headache persists for more than 7 days, an epidural 'blood patch' may be advised for relief. This procedure involves the collection of blood from your arm, which is then administered into the epidural space outside the membrane surrounding the spinal cord to seal the LP needle tract that is leaking fluid. This is effective in eliminating the headache in about 90% of people with post- spinal tap headache.

Rarer problems with an LP include:

- About 3 in 100 individuals with post-LP headache also develop double vision that can last a few days to a few weeks.
- About 3 in 100 individuals will develop temporary hearing problems or ringing in the ears lasting a few days.

Because of the risk of temporary visual blurring or headache, you should plan on having your study partner attend the procedure for transportation after the procedure, in case you are temporarily unable to drive.

#### Unforeseen Risks

You will be monitored carefully from the beginning of the procedure until the conclusion of the post-procedure rest time. The study doctor or other qualified study clinician(s) will be physically available on the CU campus if any questions arise during the lumbar puncture. The research coordinator and performing clinician will be present through the entire duration of the procedure. You will be contacted by phone approximately 1 (+/- 1) business days after the procedure to confirm your well-being and asked about any new adverse events.

#### WHAT ARE THE POSSIBLE BENEFITS OF THIS STUDY?

There are no direct benefits to participating in this lumbar puncture study. However, the information may lead to better understanding of Alzheimer's disease, how the main study drug, sargramostim, interacts with proteins, such as amyloid beta, in the brain, and how the brain responds to treatment with the study drug, sargramostim.

#### WHO IS PAYING FOR THIS STUDY?

The study is being paid for by grants from organizations like the Alzheimer's Association, the National Institutes of Health, and funds from the University of Colorado Alzheimer's and Cognition Center.

#### WILL I BE PAID FOR BEING IN THE STUDY?

To help defray your cost of participation for items such as travel costs, you will receive a \$75.00 gift card after each (optional) LP procedure, for a total maximum of \$150.00.

It is important to know that payments for participation in a study are taxable income.

#### WILL I HAVE TO PAY FOR ANYTHING?

It will not cost you anything to be in the optional lumbar puncture study.

#### IS MY PARTICIPATION VOLUNTARY?

Taking part in this optional procedure is voluntary. You have the right to choose not to take part in this optional procedure. If you choose to take part, you have the right to stop at any time. If you refuse or decide to withdraw later, you will not lose any benefits or rights to which you are entitled. You can choose not to take part in this optional procedure, and still participate in the main study.

If there are any new findings during the study that may affect whether you want to continue to take part, you will be told about them.

#### **CAN I BE REMOVED FROM THIS STUDY?**

The study doctor may decide to stop your participation without your permission if the study doctor thinks that being in the study may cause you harm, or for any other reason.

#### WHAT HAPPENS IF I AM INJURED OR HURT DURING THE STUDY?

If you have an injury while you are in this study, you should call Dr. Huntington Potter (303-724-7385) immediately. If you consider an event to be an emergency, please call 911 for emergency services.

We will arrange to get you medical care if you have an injury that is caused by this research. However, you or your insurance company will have to pay for that care.

#### WHO DO I CALL IF I HAVE QUESTIONS?

The researcher carrying out this study is Dr. Huntington Potter. You may ask any questions you have now. If you have questions, concerns, or complaints later, you may call Dr. Huntington Potter at 303-724-7385. You will be given a copy of this form to keep.

You may have questions about your rights as someone in this study. You can call the study doctors with questions. You can also call the responsible Institutional Review Board (COMIRB). You can call them at 303-724-1055.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### What happens to data collected in this study?

The data we collect will be used for this study but may also be important for future research. Your data may be used for future research or distributed to other researchers for future study without additional consent if information that identifies you is removed from the data.

#### **Certificate of Confidentiality**

This study has been issued a Certificate of Confidentiality from the federal government to help protect your privacy. The Certificate prohibits the researchers from disclosing your name, or any identifiable information, document or biospecimen from the research, with the exceptions listed below. A

certificate provides protections against disclosing research information in federal, state, or local civil, criminal, administrative, legislative or other proceedings.

These protections apply only to your research records. The protections do not apply to your medical records.

The researchers may disclose your name or identifiable information, document or biospecimen, under the following circumstances:

To those connected with the research,

If required by Federal, State or local laws,

If necessary for your medical treatment, with your consent,

For other scientific research conducted in compliance with Federal regulations,

To comply with mandated reporting, such as a possible threat to harm yourself or others, reports of child abuse, and required communicable disease reporting, or

Under other circumstances with your consent.

A Certificate of Confidentiality does not protect information you or a member of your family voluntarily release.

#### WHO WILL SEE MY RESEARCH INFORMATION?

The University of Colorado Denver | Anschutz Medical Campus (the University) and its affiliated health systems have rules to protect information about you. Federal and state laws including the Health Insurance Portability and Accountability Act (HIPAA) also protect your privacy. This part of the consent form tells you what information about you may be collected in this study and who might see or use it.

The institutions involved in this study include

- University of Colorado Denver | Anschutz Medical Campus
- University of Colorado Health

We cannot do this study without your permission to see, use and give out your information. You do not have to give us this permission. If you do not, then you may not join this study.

We will see, use and disclose your information only as described in this form and in our Notice of Privacy Practices; however, people outside the University and its affiliate hospitals may not be covered by this obligation.

We will do everything we can to maintain the confidentiality of your personal information t, but confidentiality cannot be guaranteed.

The use and disclosure of your information has no time limit. You can cancel your permission to use and disclose your information at any time by writing to the study's Sponsor, at the name and address listed below. If you do cancel your permission to use and disclose your information, your part in this study will end and no further information about you will be collected. Your cancellation would not affect information already collected in this study.

Huntington Potter, Ph.D.

Director of Alzheimer's Disease Programs Anschutz Medical Campus University of Colorado MS 8608 12700 E. 19th Ave. Aurora. CO 80045

Both the research records that identify you and the consent form signed by you may be looked at by others who have a legal right to see that information, such as:

- Federal offices such as the Food and Drug Administration (FDA), the National Institutes of Health (NIH) and the Office of Human Research Protections (OHRP) that protect research subjects like you.
- The Institutional Review Board that is responsible for overseeing this research
- The study doctor and the rest of the study team.
- Officials at the institution where the research is conducted and officials at other institutions involved in this study who are in charge of making sure that we follow all of the rules for research
- The Data Safety Monitoring Board (the committee that reviews the safety of the study).

We might talk about this research study at meetings. We might also print the results of this research study in relevant journals. But we will always keep the names and any other personally identifiable information of the research participants, like you, private.

You have the right to request access to your personal health information from the Investigator. To ensure proper evaluation of test results, your access to these study results may not be allowed until after the study is completed.

## INFORMATION ABOUT YOU THAT WILL BE SEEN, COLLECTED, USED AND DISCLOSED IN THIS STUDY:

- Name and demographic information (age, sex, ethnicity, address, phone number, etc.)
- Research test results

#### WHAT HAPPENS TO DATA AND SAMPLES) THAT ARE COLLECTED IN THIS STUDY?

Scientists at the University of Colorado Anschutz Medical Campus and the hospitals involved in this study work to find the causes and cures of disease. The data and samples collected from you during this study are important to this study and to future research. If you join this study:

- The data and samples given by you to the investigators for this research no longer belongs to you.
- Both the investigators and any sponsor of this research may study your data and samples collected from you.
- If datais or samples are in a form that identifies you, CU AMC or the hospitals involved in this study may use them for future research only with your consent or Institutional Review Board (IRB) approval.
- Any product or idea created by the researchers working on this study will not belong to you.

• There is no plan for you to receive any financial benefit from the creation, use or sale of such a product or idea.

#### AGREEMENT TO BE IN THIS OPTIONAL LUMBAR PUNCTURE STUDY AND USE MY DATA

I have read this paper about the optional lumbar puncture study or it was read to me. I understand the possible risks and benefits of the procedure. I understand and authorize the access, use and disclosure of my information as stated in this form. I know that being in this study is voluntary. I choose to be in this study: I will get a signed and dated copy of this consent form.

| Signature: | Date: |
|---------------------------------------------------------------|--------|
| Print Name: | |
| Signature Line For Legally Authorized Representative, if appl | icable |
| Legally Authorized Representative | Date |
| Print Name: | |
| Consent form explained by: | Date: |
| Print Name: | |

**PARTICIPANT**